CLINICAL TRIAL: NCT04717349
Title: Data Collection Study of Pediatric and Adolescent Gynecology Conditions
Status: Recruiting | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 200126; 20-CH-0126
Record Dates: First submitted 2021-01-20; First posted 2021-01-22 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09-10

CONDITIONS: Disorders of Sex Development (DSD); Pediatric and Adolescent Cancers of the Genital Tract; Reproductive Endocrine Conditions in Puberty; Structural Gynecologic Conditions Including Vulvar and Vaginal Conditions
Keywords: Congenital Anomalies; Disorders of sex development (DSD); Childhood and adolescence cancers; Adolescent fertility; Natural History
MeSH Terms: conditions — Disorders of Sex Development; Congenital Abnormalities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Family Members of PAG patients: Clinical evaluation of family members that would provide clinical information related to the diagnosis of a proband in future research.
- PAG patient: Pediatric and adolescent patients with gynecologic conditions.

SUMMARY:
Background:

Gynecologic conditions are those that are related to the reproductive system. They can be reproductive gland disorders or reproductive system tumors. They can also be inborn anomalies of the reproductive tract. Researchers want to gather data over time from a large group of young people with these conditions.

Objective:

To create a database about child and teenage gynecologic conditions.

Eligibility:

Participants of any age with known or suspected pediatric and adolescent gynecologic conditions, and their adult family members

Design:

Participants will be screened with a review of their medical records.

Participants may have a medical history and physical exam.

Participants will have blood drawn using a needle. The blood will be used for genetic tests.

Participants will have saliva collected. They will spit into a small plastic container. Or their spit will be absorbed from their mouth using a small sponge. The saliva will be used for genetic tests.

Participants may have samples collected from their vagina. A small cotton swab will be used to gather the samples. This procedure is optional.

If participants have a surgery related to their condition, a small tissue sample will be taken. It will be stored for future research.

Participants may complete optional surveys. These surveys ask about their physical and emotional health. They can choose not to answer any of the questions.

Researchers will collect medical data from participants standard tests. Such tests may include blood and urine tests, X-rays, nuclear medicine scans, and other tests. Data will also be collected from standard treatments they may receive.

DETAILED DESCRIPTION:
Study Description:

The overall purpose of Pediatric and Adolescent Gynecology (PAG) evaluations under this protocol is to gather information over time from a large group of patients with PAG conditions to help improve our understanding of these conditions. Our aim is to create a large database of PAG conditions in presentation and variety.

Objectives:

Primary Objective:

* Recruit a diverse population of pediatric and adult subjects with known or suspected PAG disorders in order to collect data and specimen of typical and atypical presentations of PAG disorders.
* Create a large database of PAG conditions in presentation and variety.

ELIGIBILITY:
* INCLUSION CRITERIA FOR PAG PATIENTS:

  1. Provision of signed and dated informed consent form.
  2. Stated willingness to comply with all study procedures and availability for the duration of the study.
  3. Participants with known or suspected pediatric and adolescent gynecologic conditions of any age are eligible for this protocol.

INCLUSION CRITERIA FOR PAG PATIENTS OF FAMILY MEMBERS:

1. Provision of signed and dated informed consent form.
2. Stated willingness to comply with all study procedures and availability for the duration of the study.
3. In order to be eligible to participate in this study, an individual must meet all of the following criteria: Relatives ages 18 years and older may be enrolled if clinically indicated for the diagnosis of a proband.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Any medical, physical, psychiatric, or social conditions, which, in the opinion of the investigators, would make participation in this protocol not in the best interest of the patient, will exclude participation. Patients who are critically ill, unstable, or with severe organ failure that may affect/limit the evaluation and place unsustainable demands on Clinical Center or NICHD resources will be excluded.
2. Pregnant family members

Ages: 1 Day to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Pediatric and adolescent patients with gynecologic conditions and their family members that would provide clinical information related to the diagnosis of a proband.
Sampling Method: Non-Probability Sample
Enrollment: 11000 (Estimated)
Dates: Start 2021-04-21 (Actual); Primary Completion 2039-12-02 (Estimated); Study Completion 2039-12-02 (Estimated)

PRIMARY OUTCOMES:
Recruit a diverse population of pediatric and adult subjects | Ongoing
  Recruit a diverse population of pediatric and adult subjects with known or suspected PAG disorders in order to collect evaluate the underlying natural history data and specimen of typical and atypical presentations of PAG disorders.
Create a large database of PAG conditions | Ongoing
  Create a large database of PAG conditions in presentation and variety.

CONTACTS AND LOCATIONS:
Overall Officials: Veronica Gomez-Lobo, M.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2020-CH-0126.html